CLINICAL TRIAL: NCT00494169
Title: Molecular Basis of Inherited Reproductive Disorders
Brief Title: Investigation of the Genetic Causes of Kallmann Syndrome and Reproductive Disorders
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Stephanie B. Seminara, MD, Chief, Reproductive Endocrine Unit; Professor of Medicine, Harvard Medical School; Director, Harvard Reproductive Endocrine Sciences Center, Massachusetts General Hospital
Other Study IDs: U54HD028138 (NIH)
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Hypogonadotropic Hypogonadism; Kallmann Syndrome; Puberty, Delayed; Puberty, Precocious; GnRH Deficiency
Keywords: Idiopathic Hypogonadotropic Hypogonadism; Kallmann Syndrome; Puberty; Pituitary Abnormalities; Hypothalamus; GnRH deficiency
MeSH Terms: conditions — Hypogonadism; Kallmann Syndrome; Puberty, Delayed; Puberty, Precocious; Idiopathic Hypogonadotropic Hypogonadism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — WBC are transformed into immortalized cell lines.
Oversight: Data Monitoring Committee: No

SUMMARY:
The aims of this study are: 1) to identify genes that play a role in human pubertal development and reproduction, 2) to characterize the phenotypic spectrum of patients with these gene defects, and 3) to discern the mode of inheritance for disorders caused by these gene defects. We are specifically interested in genes that cause Kallmann syndrome, idiopathic hypogonadotropic hypogonadism (IHH), precocious (early) puberty, and delayed puberty. Individuals do not have to travel to Boston to participate in this study.

DETAILED DESCRIPTION:
Overview:

Our work is divided into two main areas of investigation:

1. the discovery of new, yet-undiscovered genes for conditions of early (i.e. precocious) puberty, delayed puberty, and/or absence of pubertal development (i.e. Kallmann syndrome/hypogonadotropic hypogonadism). Identification of new genes requires either a single large family or a collection of smaller families.
2. a detailed examination of the genes already implicated in causing these conditions.

There are several other important aspects about our program:

* This analysis will detect DNA abnormalities only in those DNA segments being screened. The turnaround time to process a sample is approximately 12-24 months. We must receive a signed consent form in order to begin analysis on a blood sample.
* Our laboratory is located in Massachusetts General Hospital, Boston MA and is largely funded by the National Institutes of Health. We are a research laboratory and not a CLIA certified clinical laboratory.
* Even if a participant is the only member of his/her family affected by one of the conditions mentioned above, obtaining blood samples on other family members, including parents and siblings is often important to our work.
* It is every individual's responsibility to notify the research team he/she would like to obtain research results. Research results will be relayed to the participant's healthcare provider and must be confirmed in a clinical laboratory before being relayed to the participant or used for medical care.

Study Procedures and Risks

* You will be asked to give approximately 3-5 tablespoons of blood for this research project. There is a risk of bruising and a very small amount of bleeding associated with blood drawing.
* You will be asked to fill out a medical history checklist, indicating the presence or absence of clinical features that may be associated with abnormalities in pubertal development.
* Since absence of puberty is sometimes associated with limited or no smell ability, you may be asked to try to identify the odors in a scratch and sniff test. This will take about 15 minutes.
* Your family history can give us clues to determine how your condition was inherited. Therefore, a detailed family history, at least back to your grandparents will be obtained by a researcher.

Benefits:

There are no direct benefits to you from participation in this study. Some genes for this condition are known, other genes have yet to be discovered. If this study discovers what genes are responsible, it will help to further the understanding of this disorder. It is possible that the genetic cause of your reproductive disorder may be learned. This information can be shared with you at your request, as explained above.

When contacting us, please include in your message a description of your diagnosis, your pubertal history (age when you hit pubertal hallmarks, e.g., growth spurt; body hair; voice deepening and genital growth for men; menstruation and breast development for women) and your reproductive history.

ELIGIBILITY:
Inclusion Criteria:

* Failure to go through a normal, age-appropriate, spontaneous puberty, and abnormal hormone levels OR
* Children with abnormally early development of puberty (Precocious Puberty) OR
* Family members of these patients.

Exclusion Criteria:

* pituitary tumor
* high prolactin levels

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who
  1. fail to go through a normal, age-appropriate, spontaneous puberty, and abnormal hormone levels.
  2. have abnormally early development of puberty (Precocious Puberty)
  3. Family members of these patients.
Sampling Method: Non-Probability Sample
Enrollment: 4042 (Actual)
Dates: Start 1999-01; Primary Completion 2022-02 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Identification of DNA abnormalities | 5/2015

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie B Seminara, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Kallmann FJ, Schoenfeld WA. The genetic aspects of primary eunuchoidism. American Journal of Mental Deficiency 158:203-236, 1944.
- [Background] Franco B, Guioli S, Pragliola A, Incerti B, Bardoni B, Tonlorenzi R, Carrozzo R, Maestrini E, Pieretti M, Taillon-Miller P, Brown CJ, Willard HF, Lawrence C, Graziella Persico M, Camerino G, Ballabio A. A gene deleted in Kallmann's syndrome shares homology with neural cell adhesion and axonal path-finding molecules. Nature. 1991 Oct 10;353(6344):529-36. doi: 10.1038/353529a0. PMID 1922361
- [Background] Legouis R, Hardelin JP, Levilliers J, Claverie JM, Compain S, Wunderle V, Millasseau P, Le Paslier D, Cohen D, Caterina D, et al. The candidate gene for the X-linked Kallmann syndrome encodes a protein related to adhesion molecules. Cell. 1991 Oct 18;67(2):423-35. doi: 10.1016/0092-8674(91)90193-3. PMID 1913827
- [Background] Burris TP, Guo W, McCabe ER. The gene responsible for adrenal hypoplasia congenita, DAX-1, encodes a nuclear hormone receptor that defines a new class within the superfamily. Recent Prog Horm Res. 1996;51:241-59; discussion 259-60. PMID 8701082
- [Background] de Roux N, Young J, Misrahi M, Genet R, Chanson P, Schaison G, Milgrom E. A family with hypogonadotropic hypogonadism and mutations in the gonadotropin-releasing hormone receptor. N Engl J Med. 1997 Nov 27;337(22):1597-602. doi: 10.1056/NEJM199711273372205. No abstract available. PMID 9371856
- [Background] Layman LC, Cohen DP, Jin M, Xie J, Li Z, Reindollar RH, Bolbolan S, Bick DP, Sherins RR, Duck LW, Musgrove LC, Sellers JC, Neill JD. Mutations in gonadotropin-releasing hormone receptor gene cause hypogonadotropic hypogonadism. Nat Genet. 1998 Jan;18(1):14-5. doi: 10.1038/ng0198-14. No abstract available. PMID 9425890
- [Background] Crowley WF Jr, Pitteloud N, Seminara S. New genes controlling human reproduction and how you find them. Trans Am Clin Climatol Assoc. 2008;119:29-37; discussion 37-8. PMID 18596868
- [Background] Balasubramanian R, Plummer L, Sidis Y, Pitteloud N, Martin C, Zhou QY, Crowley WF Jr. The puzzles of the prokineticin 2 pathway in human reproduction. Mol Cell Endocrinol. 2011 Oct 22;346(1-2):44-50. doi: 10.1016/j.mce.2011.05.040. Epub 2011 Jun 1. PMID 21664414
- [Background] Au MG, Crowley WF Jr, Buck CL. Genetic counseling for isolated GnRH deficiency. Mol Cell Endocrinol. 2011 Oct 22;346(1-2):102-9. doi: 10.1016/j.mce.2011.05.041. Epub 2011 Jun 1. PMID 21664415
- [Result] Pitteloud N, Meysing A, Quinton R, Acierno JS Jr, Dwyer AA, Plummer L, Fliers E, Boepple P, Hayes F, Seminara S, Hughes VA, Ma J, Bouloux P, Mohammadi M, Crowley WF Jr. Mutations in fibroblast growth factor receptor 1 cause Kallmann syndrome with a wide spectrum of reproductive phenotypes. Mol Cell Endocrinol. 2006 Jul 25;254-255:60-9. doi: 10.1016/j.mce.2006.04.021. Epub 2006 Jun 9. PMID 16764984
- [Result] Pallais JC, Bo-Abbas Y, Pitteloud N, Crowley WF Jr, Seminara SB. Neuroendocrine, gonadal, placental, and obstetric phenotypes in patients with IHH and mutations in the G-protein coupled receptor, GPR54. Mol Cell Endocrinol. 2006 Jul 25;254-255:70-7. doi: 10.1016/j.mce.2006.04.019. Epub 2006 Jun 6. PMID 16757106
- [Result] Pitteloud N, Acierno JS Jr, Meysing A, Eliseenkova AV, Ma J, Ibrahimi OA, Metzger DL, Hayes FJ, Dwyer AA, Hughes VA, Yialamas M, Hall JE, Grant E, Mohammadi M, Crowley WF Jr. Mutations in fibroblast growth factor receptor 1 cause both Kallmann syndrome and normosmic idiopathic hypogonadotropic hypogonadism. Proc Natl Acad Sci U S A. 2006 Apr 18;103(16):6281-6. doi: 10.1073/pnas.0600962103. Epub 2006 Apr 10. PMID 16606836
- [Result] Pitteloud N, Acierno JS Jr, Meysing AU, Dwyer AA, Hayes FJ, Crowley WF Jr. Reversible kallmann syndrome, delayed puberty, and isolated anosmia occurring in a single family with a mutation in the fibroblast growth factor receptor 1 gene. J Clin Endocrinol Metab. 2005 Mar;90(3):1317-22. doi: 10.1210/jc.2004-1361. Epub 2004 Dec 21. PMID 15613419
- [Result] Teles MG, Bianco SD, Brito VN, Trarbach EB, Kuohung W, Xu S, Seminara SB, Mendonca BB, Kaiser UB, Latronico AC. A GPR54-activating mutation in a patient with central precocious puberty. N Engl J Med. 2008 Feb 14;358(7):709-15. doi: 10.1056/NEJMoa073443. PMID 18272894
- [Result] Cerrato F, Seminara SB. Human genetics of GPR54. Rev Endocr Metab Disord. 2007 Mar;8(1):47-55. doi: 10.1007/s11154-007-9027-3. PMID 17334928
- [Result] Pitteloud N, Zhang C, Pignatelli D, Li JD, Raivio T, Cole LW, Plummer L, Jacobson-Dickman EE, Mellon PL, Zhou QY, Crowley WF Jr. Loss-of-function mutation in the prokineticin 2 gene causes Kallmann syndrome and normosmic idiopathic hypogonadotropic hypogonadism. Proc Natl Acad Sci U S A. 2007 Oct 30;104(44):17447-52. doi: 10.1073/pnas.0707173104. Epub 2007 Oct 24. PMID 17959774
- [Result] Cerrato F, Shagoury J, Kralickova M, Dwyer A, Falardeau J, Ozata M, Van Vliet G, Bouloux P, Hall JE, Hayes FJ, Pitteloud N, Martin KA, Welt C, Seminara SB. Coding sequence analysis of GNRHR and GPR54 in patients with congenital and adult-onset forms of hypogonadotropic hypogonadism. Eur J Endocrinol. 2006 Nov;155 Suppl 1:S3-S10. doi: 10.1530/eje.1.02235. PMID 17074994
- [Result] Bo-Abbas Y, Acierno JS Jr, Shagoury JK, Crowley WF Jr, Seminara SB. Autosomal recessive idiopathic hypogonadotropic hypogonadism: genetic analysis excludes mutations in the gonadotropin-releasing hormone (GnRH) and GnRH receptor genes. J Clin Endocrinol Metab. 2003 Jun;88(6):2730-7. doi: 10.1210/jc.2002-021948. PMID 12788881
- [Result] Seminara SB, Messager S, Chatzidaki EE, Thresher RR, Acierno JS Jr, Shagoury JK, Bo-Abbas Y, Kuohung W, Schwinof KM, Hendrick AG, Zahn D, Dixon J, Kaiser UB, Slaugenhaupt SA, Gusella JF, O'Rahilly S, Carlton MB, Crowley WF Jr, Aparicio SA, Colledge WH. The GPR54 gene as a regulator of puberty. N Engl J Med. 2003 Oct 23;349(17):1614-27. doi: 10.1056/NEJMoa035322. PMID 14573733
- [Result] Jongmans MC, van Ravenswaaij-Arts CM, Pitteloud N, Ogata T, Sato N, Claahsen-van der Grinten HL, van der Donk K, Seminara S, Bergman JE, Brunner HG, Crowley WF Jr, Hoefsloot LH. CHD7 mutations in patients initially diagnosed with Kallmann syndrome--the clinical overlap with CHARGE syndrome. Clin Genet. 2009 Jan;75(1):65-71. doi: 10.1111/j.1399-0004.2008.01107.x. Epub 2008 Nov 17. PMID 19021638
- [Result] Chan YM, de Guillebon A, Lang-Muritano M, Plummer L, Cerrato F, Tsiaras S, Gaspert A, Lavoie HB, Wu CH, Crowley WF Jr, Amory JK, Pitteloud N, Seminara SB. GNRH1 mutations in patients with idiopathic hypogonadotropic hypogonadism. Proc Natl Acad Sci U S A. 2009 Jul 14;106(28):11703-8. doi: 10.1073/pnas.0903449106. Epub 2009 Jun 30. PMID 19567835
- [Result] Gianetti E, Tusset C, Noel SD, Au MG, Dwyer AA, Hughes VA, Abreu AP, Carroll J, Trarbach E, Silveira LF, Costa EM, de Mendonca BB, de Castro M, Lofrano A, Hall JE, Bolu E, Ozata M, Quinton R, Amory JK, Stewart SE, Arlt W, Cole TR, Crowley WF, Kaiser UB, Latronico AC, Seminara SB. TAC3/TACR3 mutations reveal preferential activation of gonadotropin-releasing hormone release by neurokinin B in neonatal life followed by reversal in adulthood. J Clin Endocrinol Metab. 2010 Jun;95(6):2857-67. doi: 10.1210/jc.2009-2320. Epub 2010 Mar 23. PMID 20332248
- [Result] Sykiotis GP, Pitteloud N, Seminara SB, Kaiser UB, Crowley WF Jr. Deciphering genetic disease in the genomic era: the model of GnRH deficiency. Sci Transl Med. 2010 May 19;2(32):32rv2. doi: 10.1126/scitranslmed.3000288. PMID 20484732
- [Result] Sykiotis GP, Plummer L, Hughes VA, Au M, Durrani S, Nayak-Young S, Dwyer AA, Quinton R, Hall JE, Gusella JF, Seminara SB, Crowley WF Jr, Pitteloud N. Oligogenic basis of isolated gonadotropin-releasing hormone deficiency. Proc Natl Acad Sci U S A. 2010 Aug 24;107(34):15140-4. doi: 10.1073/pnas.1009622107. Epub 2010 Aug 9. PMID 20696889
- [Result] Martin C, Balasubramanian R, Dwyer AA, Au MG, Sidis Y, Kaiser UB, Seminara SB, Pitteloud N, Zhou QY, Crowley WF Jr. The role of the prokineticin 2 pathway in human reproduction: evidence from the study of human and murine gene mutations. Endocr Rev. 2011 Apr;32(2):225-46. doi: 10.1210/er.2010-0007. Epub 2010 Oct 29. PMID 21037178
- [Result] Shaw ND, Seminara SB, Welt CK, Au MG, Plummer L, Hughes VA, Dwyer AA, Martin KA, Quinton R, Mericq V, Merino PM, Gusella JF, Crowley WF Jr, Pitteloud N, Hall JE. Expanding the phenotype and genotype of female GnRH deficiency. J Clin Endocrinol Metab. 2011 Mar;96(3):E566-76. doi: 10.1210/jc.2010-2292. Epub 2011 Jan 5. PMID 21209029
- [Result] Caronia LM, Martin C, Welt CK, Sykiotis GP, Quinton R, Thambundit A, Avbelj M, Dhruvakumar S, Plummer L, Hughes VA, Seminara SB, Boepple PA, Sidis Y, Crowley WF Jr, Martin KA, Hall JE, Pitteloud N. A genetic basis for functional hypothalamic amenorrhea. N Engl J Med. 2011 Jan 20;364(3):215-25. doi: 10.1056/NEJMoa0911064. PMID 21247312
- [Result] Tornberg J, Sykiotis GP, Keefe K, Plummer L, Hoang X, Hall JE, Quinton R, Seminara SB, Hughes V, Van Vliet G, Van Uum S, Crowley WF, Habuchi H, Kimata K, Pitteloud N, Bulow HE. Heparan sulfate 6-O-sulfotransferase 1, a gene involved in extracellular sugar modifications, is mutated in patients with idiopathic hypogonadotrophic hypogonadism. Proc Natl Acad Sci U S A. 2011 Jul 12;108(28):11524-9. doi: 10.1073/pnas.1102284108. Epub 2011 Jun 23. PMID 21700882
- [Result] Lewkowitz-Shpuntoff HM, Hughes VA, Plummer L, Au MG, Doty RL, Seminara SB, Chan YM, Pitteloud N, Crowley WF Jr, Balasubramanian R. Olfactory phenotypic spectrum in idiopathic hypogonadotropic hypogonadism: pathophysiological and genetic implications. J Clin Endocrinol Metab. 2012 Jan;97(1):E136-44. doi: 10.1210/jc.2011-2041. Epub 2011 Nov 9. PMID 22072740
- [Result] Gianetti E, Hall JE, Au MG, Kaiser UB, Quinton R, Stewart JA, Metzger DL, Pitteloud N, Mericq V, Merino PM, Levitsky LL, Izatt L, Lang-Muritano M, Fujimoto VY, Dluhy RG, Chase ML, Crowley WF Jr, Plummer L, Seminara SB. When genetic load does not correlate with phenotypic spectrum: lessons from the GnRH receptor (GNRHR). J Clin Endocrinol Metab. 2012 Sep;97(9):E1798-807. doi: 10.1210/jc.2012-1264. Epub 2012 Jun 28. PMID 22745237
- [Result] Avbelj Stefanija M, Jeanpierre M, Sykiotis GP, Young J, Quinton R, Abreu AP, Plummer L, Au MG, Balasubramanian R, Dwyer AA, Florez JC, Cheetham T, Pearce SH, Purushothaman R, Schinzel A, Pugeat M, Jacobson-Dickman EE, Ten S, Latronico AC, Gusella JF, Dode C, Crowley WF Jr, Pitteloud N. An ancient founder mutation in PROKR2 impairs human reproduction. Hum Mol Genet. 2012 Oct 1;21(19):4314-24. doi: 10.1093/hmg/dds264. Epub 2012 Jul 5. PMID 22773735
- [Result] Chew S, Balasubramanian R, Chan WM, Kang PB, Andrews C, Webb BD, MacKinnon SE, Oystreck DT, Rankin J, Crawford TO, Geraghty M, Pomeroy SL, Crowley WF Jr, Jabs EW, Hunter DG, Grant PE, Engle EC. A novel syndrome caused by the E410K amino acid substitution in the neuronal beta-tubulin isotype 3. Brain. 2013 Feb;136(Pt 2):522-35. doi: 10.1093/brain/aws345. Epub 2013 Jan 31. PMID 23378218
- [Result] Costa-Barbosa FA, Balasubramanian R, Keefe KW, Shaw ND, Al-Tassan N, Plummer L, Dwyer AA, Buck CL, Choi JH, Seminara SB, Quinton R, Monies D, Meyer B, Hall JE, Pitteloud N, Crowley WF Jr. Prioritizing genetic testing in patients with Kallmann syndrome using clinical phenotypes. J Clin Endocrinol Metab. 2013 May;98(5):E943-53. doi: 10.1210/jc.2012-4116. Epub 2013 Mar 26. PMID 23533228
- [Result] Miraoui H, Dwyer AA, Sykiotis GP, Plummer L, Chung W, Feng B, Beenken A, Clarke J, Pers TH, Dworzynski P, Keefe K, Niedziela M, Raivio T, Crowley WF Jr, Seminara SB, Quinton R, Hughes VA, Kumanov P, Young J, Yialamas MA, Hall JE, Van Vliet G, Chanoine JP, Rubenstein J, Mohammadi M, Tsai PS, Sidis Y, Lage K, Pitteloud N. Mutations in FGF17, IL17RD, DUSP6, SPRY4, and FLRT3 are identified in individuals with congenital hypogonadotropic hypogonadism. Am J Hum Genet. 2013 May 2;92(5):725-43. doi: 10.1016/j.ajhg.2013.04.008. PMID 23643382
- [Result] Salian-Mehta S, Xu M, Knox AJ, Plummer L, Slavov D, Taylor M, Bevers S, Hodges RS, Crowley WF Jr, Wierman ME. Functional consequences of AXL sequence variants in hypogonadotropic hypogonadism. J Clin Endocrinol Metab. 2014 Apr;99(4):1452-60. doi: 10.1210/jc.2013-3426. Epub 2014 Jan 29. PMID 24476074
- [Derived] Delaney A, Burkholder AB, Lavender CA, Plummer L, Mericq V, Merino PM, Quinton R, Lewis KL, Meader BN, Albano A, Shaw ND, Welt CK, Martin KA, Seminara SB, Biesecker LG, Bailey-Wilson JE, Hall JE. Increased Burden of Rare Sequence Variants in GnRH-Associated Genes in Women With Hypothalamic Amenorrhea. J Clin Endocrinol Metab. 2021 Mar 8;106(3):e1441-e1452. doi: 10.1210/clinem/dgaa609. PMID 32870266
- [Derived] Lippincott MF, Leon S, Chan YM, Fergani C, Talbi R, Farooqi IS, Jones CM, Arlt W, Stewart SE, Cole TR, Terasawa E, Hall JE, Shaw ND, Navarro VM, Seminara SB. Hypothalamic Reproductive Endocrine Pulse Generator Activity Independent of Neurokinin B and Dynorphin Signaling. J Clin Endocrinol Metab. 2019 Oct 1;104(10):4304-4318. doi: 10.1210/jc.2019-00146. PMID 31132118
- [Derived] Raivio T, Avbelj M, McCabe MJ, Romero CJ, Dwyer AA, Tommiska J, Sykiotis GP, Gregory LC, Diaczok D, Tziaferi V, Elting MW, Padidela R, Plummer L, Martin C, Feng B, Zhang C, Zhou QY, Chen H, Mohammadi M, Quinton R, Sidis Y, Radovick S, Dattani MT, Pitteloud N. Genetic overlap in Kallmann syndrome, combined pituitary hormone deficiency, and septo-optic dysplasia. J Clin Endocrinol Metab. 2012 Apr;97(4):E694-9. doi: 10.1210/jc.2011-2938. Epub 2012 Feb 8. PMID 22319038